CLINICAL TRIAL: NCT04056104
Title: Improving Critical Congenital Heart Disease Screening With Addition of Perfusion Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1386243; 5KL2TR001859-04 (NIH); R21HD099239-01 (NIH)
Record Dates: First submitted 2019-07-22; First posted 2019-08-14 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Oxygen Saturation

STUDY DESIGN:
Intervention Model Description: Non-invasive measurements of oxygenation and perfusion will be measured with pulse oximeters
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SpO2 and PIx Measurement (Experimental): Non-invasive measurements of oxygenation (SpO2) and perfusion (PIx) will be measured with pulse oximeters
  Interventions: Diagnostic Test: SpO2 and PIx Measurement

INTERVENTIONS:
Diagnostic Test: SpO2 and PIx Measurement — Right upper and any lower extremity oxygen saturation (SpO2) and perfusion index (PIx) will be measured

SUMMARY:
The purpose of this research is to evaluate and create a new clinical prediction model for CCHD screening that combines non-invasive measurements of oxygenation and perfusion.

DETAILED DESCRIPTION:
This study will create and test an enhanced critical congenital heart defect (CCHD) screen that combines non-invasive measurements of oxygenation and perfusion in two ways. The first will use current equipment without automated interpretation and the second will require additional software/device but will automate the interpretation. To work towards development of those two algorithms in this stage of the study, the study team will download oxygen saturation (SpO2) and perfusion index (PIx) measurements from newborns with and without congenital heart disease (CHD) and apply statistical tests to the data afterwards to identify parameters to include in the newly developed screening algorithms. The overall objective is to create an automated screening algorithm to improve acyanotic CCHD detection, preventing morbidity and mortality associated with diagnoses missed by SpO2 screening. The central hypothesis is that the addition of non-invasive perfusion measurements to SpO2 will be superior to SpO2-alone screening for detection of acyanotic CCHD. The data collected during this study will be used to develop the two algorithms and the algorithms will be compared to the standard of care using statistical tests on the data after the fact (k-fold validation). The newly developed algorithms will not be tested in-situ on patients during this study.

ELIGIBILITY:
Inclusion Criteria:

* Age < 22 days
* and either: a) asymptomatic newborn undergoing SpO2 screening for CCHD, or 2b) newborn prenatally or postnatally diagnosed/suspected with CHD.

Exclusion Criteria:

* For Controls: Echocardiogram completed prior to enrollment as the newborn would then no longer be considered "asymptomatic undergoing SpO2 screening for CCHD"
* For Newborns with confirmed/suspected CHD: a) Patent ductus arteriosus and/or atrial septal defect/patent foramen ovale without other defects, b) Corrective cardiac surgical or catheter intervention performed before enrollment or c) Current infusions of vasoactive medications other than prostaglandin therapy.

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 543 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristics (AUROC) of critical congenital heart defect (CCHD) screening algorithm for CCHD with systemic obstruction from coarctation of the aorta or interrupted aortic arch | At enrollment
  A CCHD screening algorithm will be created by simultaneously measuring oxygen saturation, perfusion index, and pulse oximetry waveform analysis from right upper and any lower extremity in newborns with and without CHD. Investigators will use cross-validation to test the newly developed algorithms and estimate AUROC for the specified types of heart defects. For purposes of defining primary and secondary criterion variables, the CHD will be considered present or absent at enrollment when the infant is less than 22 days of age according to the latest diagnostic assessment available for the infant (echocardiogram and/or physical examination). Because some CHDs can be diagnosed at later dates despite earlier negative diagnostic evaluations, investigators will reconfirm the presence or absence of the outcome at a minimum of 6 weeks of age for all patients except those who die or are lost to follow-up.

SECONDARY OUTCOMES:
AUROC of CCHD screening algorithm for any critical congenital heart defect (CCHD) | At 30 days of life
  AUROC of CCHD screening algorithm for any critical congenital heart defect (CCHD). CCHD will be defined as an anatomical heart defect that requires surgical or catheter-based corrective/palliative procedure in the first 30 days after birth
AUROC of CCHD screening algorithm for critical congenital heart defect (CCHD) with any systemic obstruction | At enrollment
  AUROC of CCHD screening algorithm for critical congenital heart defect (CCHD) with any systemic obstruction
AUROC of CCHD screening algorithm for any congenital heart defect (CHD) | At enrollment
  AUROC of CCHD screening algorithm for any congenital heart defect (CHD). CHD will be defined as any anatomical heart with the exception of isolated patent ductus arteriosus and/or atrial septal defect/patent foramen ovale

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Sutter Institute for Medical Research, Sacramento, California
  - University of California-Davis, Sacramento, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Northwell Health, New Hyde Park, New York
  - University of Utah/Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siefkes H, Oliveira LC, Koppel R, Hogan W, Garg M, Manalo E, Cresalia N, Lai Z, Tancredi D, Lakshminrusimha S, Chuah CN. Machine Learning-Based Critical Congenital Heart Disease Screening Using Dual-Site Pulse Oximetry Measurements. J Am Heart Assoc. 2024 Jun 18;13(12):e033786. doi: 10.1161/JAHA.123.033786. Epub 2024 Jun 15. PMID 38879455